CLINICAL TRIAL: NCT01545362
Title: The Effect of Preop Nutritional Status on Outcomes of Staged Bilateral Total Knee Replacements Performed Within One Week
Brief Title: Effect of Preop Nutritional Status on Outcomes of Staged Bilateral Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Heekin Orthopedic Research Institute (Other)
Responsible Party: Principal Investigator, R. David Heekin, MD, Principal Investigator, Heekin Orthopedic Research Institute
Other Study IDs: 2010-004
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Staged bilateral total knee arthroplasty: Patients that have bilateral total knee arthroplasty staged within one week
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Total knee arthroplasty

SUMMARY:
To determine if preop nutritional status is an indicator for outcomes of bilateral staged total knee arthroplasty. The investigators expect that patients having staged bilateral total knee arthroplasty with the second procedure performed within one week of the first and have a total lymphocyte count >1500 per cubic millimeter and serum albumin level >35 grams per liter will have the same or less complications and shorter length of stay than those with lower lymphocyte count and albumin level.

DETAILED DESCRIPTION:
Association of malnutrition with postoperative complications after TKA has been reported in the form of increased rate of periprosthetic infection, longer hospital stay, etc. Reduced serum albumin and total lymphocyte count are commonly used to define malnutrition.

The goal was to evaluate the impact of the nutritional status on the outcomes of primary staged bilateral TKAs performed one-week apart during two separate hospitalizations.

Fifty consecutive patients with mean age of 67 years, mean BMI of 28.9 and 2.3 mean ASA score were followed for one year.

Prior to the first surgery 32% had a TLC <1500 cells/mm3 and 84% had a SA <3.5 g/dL. Before the second surgery 62% had a reduced TLC and all but one had a reduced SA.

Nine patients had a total of 12 perioperative blood transfusions (2 after the first surgery and 10 after the second surgery). The average length of stay was 3 days after each TKA.

None of the patients with the lowest TLC or SA before the first or the second stage had a revision.

Bilateral TKAs performed seven days apart in two separate hospitalizations is a safe and practical approach for qualified patients. The postoperative course was similar after each surgery. The preoperative nutritional status defined by TLC and SA did not influence the postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or non-pregnant female over the age of 21.
* Patient requires a bilateral staged knee arthroplasty (within 7 days)
* Patient has signed and dated an IRB approved consent form.
* Patient is able and willing to participate in the study according to the protocol for the full length of expected term of follow-up, and to follow their physician's directions.
* Patient has failed to respond to conservative treatment modalities.

Exclusion Criteria:

* Patient's bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prosthesis.
* Patient is a prisoner.
* Surgery on the second side cancelled or delayed past 7 days by patient request subject will be terminated from the study.
* BMI >35

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort selected from patients in orthopaedic clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Blood loss until drain is pulled | postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: R. David Heekin, M.D., Principal Investigator — Heekin Institute for Orthopedic Research
Locations (1):
- Heekin Orthopedic Specialists, Jacksonville, Florida, United States